CLINICAL TRIAL: NCT01701739
Title: An Open-label, Two-period Fixed-sequence Study to Investigate the Effect of Multiple Doses of Aleglitazar on a Single Dose of Digoxin in Healthy Subjects
Brief Title: A Pharmacokinetics Study of Aleglitazar in Combination With Digoxin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP25562; 2012-002269-36 (EudraCT Number)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — aleglitazar; Digoxin

ARMS (1):
- aleglitazar / digoxin (Experimental)
  Interventions: Drug: aleglitazar; Drug: digoxin

INTERVENTIONS:
Drug: aleglitazar — Multiple doses of aleglitazar
Drug: digoxin — Single dose of digoxin

SUMMARY:
This open-label, two-period, fixed-sequence study will investigate the pharmacokinetics and safety of multiple doses of aleglitazar on a single dose of digoxin in healthy volunteers. In period 1, volunteers will receive a single dose of digoxin, in period 2 volunteers will receive multiple doses of aleglitazar and a single dose of digoxin. The anticipated time on study treatment is one month.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18-55 years of age, inclusive
* Body mass index (BMI) between 18.0 and 30.0 kg/m2 inclusive.
* Females must be either surgically sterile or post-menopausal for at least one year or, if they are of child-bearing potential, must use two acceptable methods of contracepetion
* Volunteer normally drinks no more than three cups of coffee/tea/caffeinated soft drinks per day and is willing to stop drinking coffee/tea/caffeinated soft drinks during the study

Exclusion Criteria:

* Any clinically relevant abnormal laboratory test results at screening or on Day -1
* Has taken any prescribed or herbal/over the counter medication within 2 weeks prior to the first dosing
* A history of clinically significant gastro-intestinal, cardiovascular, musculoskeletal, endocrine, hematological, psychiatric, renal, hepatic, bronchopulmonary or neurological conditions or lipid metabolism disorders.
* Infection with human immunodeficiency virus (HIV), hepatitis B, hepatitis C
* An average alcohol intake of more than 14 units per week
* A known permanent or unexplained elevation of serum transaminases > 1.5 times the upper limit of normal
* A positive screen for drugs of abuse
* Acute infection requiring treatment within 4 weeks prior to screening
* Diagnosed or treated malignancy within the past 5 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration time curve | Approximately 1 month
Pharmacokinetics: maximum plasma concentration | Approximately 1 month

SECONDARY OUTCOMES:
Pharmacokinetics: Elimination half-life | Approximately 1 month
Pharmacokinetics: Time to maximum plasma concentration | Approximately 1 month
Pharmacokinetics: Renal clearance | Approximately 1 month
Pharmacokinetics: Apparent volume of distribution | Approximately 1 month
Pharmacokinetics: Apparent clearance | Approximately 1 month
Pharmacokinetics: Amount excreted in the urine | Approximately 1 month
Pharmacokinetics: Fraction of drug excreted in urine | Approximately 1 month
Safety: Incidence of adverse events | Approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Manchester, United Kingdom